CLINICAL TRIAL: NCT06565988
Title: A Post-market-clinical Follow-up Investigation of Safety and Performance of Decoria® Voluma
Brief Title: A Post-market-clinical Follow-up Investigation of Safety and Performance by Decoria® Voluma
Acronym: DAG-VOL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bohus Biotech AB (Industry)
Collaborators: Key2Compliance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIV-24-03-046500
Record Dates: First submitted 2024-08-16; First posted 2024-08-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2024-11

CONDITIONS: Midface Volume Deficit
Keywords: tissue augmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Investigational Medical Device (Other): All eligable subjects desiring correction of cheek volume will receive intradermal injection of Decoria Voluma on either one or both sides of the face.
  Interventions: Device: Decoria Voluma

INTERVENTIONS:
Device: Decoria Voluma — Decoria® Voluma medical device is a sterile, single use Hyaloronic acid based dermal filler intended for aesthetic use, provided in the form of a nonpyrogenic, viscoelastic gel. It is composed of highly purified sodium hyaluronate of high molecular weight, dissolved in a physiological buffer at pH 6.0-7.5. The sodium hyaluronate is derived from microbial fermentation and is stabilized by crosslinking with the chemical agent BDDE (1,4 Butanediol Diglycidyl Ether).
  Decoria® Voluma dermal fillers are injected into dermal tissue for the correction of midface volume deficit by tissue augmentation in cheek region, supporting overlying tissue to shape facial contours to desired level of correction. This is possible due to the capacity of HA to attract and bind large amounts of water, forming a viscous gel.
  Appropriate injection volume for the cheek region(s) will be determined by the Treating investigator according to IFU.

SUMMARY:
A post-market-clinical follow-up investigation of safety and performance of Decoria® Voluma by the correction of midface volume deficit by tissue augmentation in cheek region.

DETAILED DESCRIPTION:
This will be a post-market, open-label, prospective, interventional, confirmatory, evaluator-blinded, multi- centre, clinical investigation to confirm the clinical safety and performance profile of Decoria® Voluma for the correction of midface volume deficit by tissue augmentation in cheek region.

Subjects desiring correction of cheek volume at the participating sites will be asked to participate in the clinical investigation. According to the national legislation, all subjects must have a consultation with the respective clinic and receive both oral and written information at least 48 hours prior to treatment with fillers, as to allow for sufficient reflection time.

If the subject decides to participate, the subject will receive treatment on Day 0 (Visit 1). At 1 month visit (Visit 2) an optional touch-up may be given as well as assessments performed. All subjects will be followed for 6 months with follow-up and assessments either by physical visits to a clinic (Visit 2 and Visit 4) or by phone call (Visit 3).

A total of 4 visits (including screening Visit 0) at the site are planned for each subject.

Standardized facial photography will be taken prior to and after treatment during Visit 1 and during each follow-up visit at the clinic (Visit 2 and 4), for evaluation according to GAIS grading and for the exploratory instrumental evaluation of cheek volume. GAIS will be used for blinded investigator assessment, treating investigator assessment and patient satisfaction.

Numeric Pain Rating Scale (NRS) at each visit involving an injection (Visit 1 and Visit 2- optional touch up) will be used to measure pain.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years, males and females.
2. Able and willing to give written informed consent for participation in the investigation.
3. Treating investigator considers the subject's cheeks amenable to an improvement of at least 1 grade on the GAIS. At least one side of face should either have a potential to enhance cheek volume or have moderate to severe cheek volume deficit. The grades do not have to be the same on both sides.
4. Ability to follow study instructions and likely to complete all required visits.

Exclusion Criteria:

1. Pregnant or lactating females.
2. Any previous hypersensitivity reaction to any constituent of the Investigational medical device (IMD) or to local anaesthetic products.
3. Any corrective procedures performed or planned in the midface region (e.g., silicone implants, permanent fillers, absorbable and non-absorbable sutures, laser therapy, dermabrasion, dental implants) that may confound the evaluation of safety and performance of the IMD.
4. Any other intradermal injection, such as semi-permanent fillers or botulinum toxin (no complications are allowed), received in the same injection area within 12 months of the Treatment visit (Visit 1) that may confound the evaluation of safety and performance of the IMD.
5. Has an ongoing episode/relapse, recently diagnosed or newly started medication of an autoimmune disease, as judged by the investigator.
6. Has any chronic or acute skin disease or inflammation (such as pimples, rashes or hives) within or close to the treatment area.
7. Has any treatments (thrombolytics, anticoagulants) or disease related to the coagulation system.
8. Subjects that have taken any type of vaccine within two weeks prior injection with the IMD.
9. Patients receiving interferon and ribavirin treatment.
10. Features that may interfere with the visual assessment such as recent cosmetic treatment,scarring, abscess, piercing or tattoo.
11. Participation in a clinical investigation that may affect the safety or performance of this investigation, as judged by the Principal Investigator, or authorized designee.
12. Employees of the study site or the sponsor directly involved with the conduct of the investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint | From pre-intervention baseline, to 6 months post-treatment
  The primary efficacy endpoint is the blinded evaluator assessment of improvement using the Global Aesthetic Improvement Scale (GAIS). GAIS is a comparative scale, based on assessment of change since before pre-intervention, which ranges from score 1 (exceptionally improved), 2 (much improved), 3 (improved), 4 (no change) to 5 (worse). The blinded evaluator will compare the pre-intervention face to post-intervention face and assign the level of improvement in cheek volume according to the GAIS grading. Each side of the face (left and right) will be assessed independently.
Primary safety endpoint | Baseline to end of study (6 months)
  The primary safety endpoint is to assess the safety of Decoria® Voluma, evaluated by the incidence, intensity, duration, and time of onset of related AEs, including injection site reactions, collected during the study duration.

SECONDARY OUTCOMES:
Secondary endpoint | Baseline (visit 1) and (visit 2) (30 days post baseline)
  1. Pain will be measured by numerical scale Numeric Pain Rating Scale (NRS) (11-point verbal score completed for each target region treated) for each visit involving an injection.
Secondary endpoint | 30 days and 180 days post treatment
  2. GAIS score at 1- and 6-months post-treatment, as assessed by the treating investigator.
Secondary endpoint | 30 days and 180 days post treatment
  3. GAIS score at 1- and 6-months post-treatment, as assessed by the subject.
Secondary endpoint | Baseline (visit 1) and (visit 2) (30 days post baseline)
  4. Treatment-related adverse events and injection site reactions reported after touch-up should be similar to those reported after initial treatment.
Secondary endpoint | Baseline, 30 days and 180 days post treatment
  5. Change in cheek volume compared to baseline will be measured after treatment, as well as at
  1- month and 6- months post-treatment visits.

CONTACTS AND LOCATIONS:
Overall Officials: Lucian Grema, M.D, Principal Investigator — Florakliniken, Stockholm, Sweden
Locations (7):
- Sweden (7):
  - Inskinity, Gothenburg
  - Göteborgs Laser & Estetik, Gothenburg
  - Svenska Hudkliniker, Karlstad
  - Inskinity, Stockholm
  - Florakliniken, Stockholm
  - The Faculty, Stockholm
  - Svenska Hudkliniker, Stockholm